CLINICAL TRIAL: NCT04959357
Title: The Evaluation of Left Ventricular Systolic Function in Different Types of Ischemic Heart Disease by Two-dimensional Speckle-tracking Echocardiography
Brief Title: The Evaluation of Left Ventricular Systolic Function in Different Types of Ischemic Heart Disease
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 048-01
Record Dates: First submitted 2021-06-27; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Coronary Microvascular Dysfunction; Obstructive Coronary Heart Disease
Keywords: two-dimensional speckle tracking imaging; strain; coronary microvascular dysfunction
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (3):
- coronary microvascular dysfunction group
  Interventions: Diagnostic Test: Two dimensional speckle tracking imaging
- obstructive coronary artery disease
  Interventions: Diagnostic Test: Two dimensional speckle tracking imaging
- control group
  Interventions: Diagnostic Test: Two dimensional speckle tracking imaging

INTERVENTIONS:
Diagnostic Test: Two dimensional speckle tracking imaging — lobal longitudinal strain and strain rate, subendocardial LS and subepicardial LS were quantified by two dimensional speckle tracking imaging

SUMMARY:
The study was designed to evaluate the left ventricular longitudinal strain and strain rate assessed by 2D-STI in patients with coronary microvascular dysfunction (CMD) or obstructive coronary artery disease (CAD) , to investigate the effect of different types of ischemic heart disease on the LV systolic function, and to explore the value of LS on the diagnosis of coronary microvascular dysfunction.

DETAILED DESCRIPTION:
A total of 175 patients with chest pain, without wall motion abnormality and without significant coronary artery stenosis (<50%) assessed by coronary angiography or coronary computed tomography were enrolled from July 2011 to December 2017. Coronary flow reserve (CFR) of these patients were detected by transthoracic Doppler echocardiography. The patients were divided into coronary microvascular dysfunction group ( CFR≤2.5, n=67) and control group (CFR>2.5, n=108). At the same time, 67 age-matched patients with any major coronary arteries stenosis≥50% and without wall motion abnormality were involved into the obstructive coronary artery disease group. Parameters of global longitudinal strain (LS) and strain rate, subendocardial LS and subepicardial LS were quantified by 2D-STI, the differences of these parameters among three groups were analyzed，correlation analysis、univariate and multivariate analysis and receiver operating characteristic curve were used.

ELIGIBILITY:
Inclusion Criteria:

* age from 18-85 years

Exclusion Criteria:

* patients with history of myocardial infarction or abnormal wall motion suggested by conventional echocardiography
* patients with acute heart failure, chronic heart failure or LVEF values less than 50%
* patients with congenital heart disease, severe valvular disease, severe bradycardia, high atrioventricular block and atrial fibrillation
* patients who did not store ultrasound images or whose ultrasound images were unclear
* patients who had incomplete clinical data

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 242 patients were enrolled, including 102 males (42.1%) and 140 females (57.9%). Their ages ranged from 44 to 81 years, with an average age of (62.6 + 8.3) years.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
global longitudinal strain | 15/3/2018-30/12/2018
  global longitudinal strain of CMD group and obstructive CAD group

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhaoping, professor, Study Chair — Peking University Third Hospital
Locations (1):
- Department of Cardiology, Peking University Third Hospital, NHC Key Laboratory of Cardiovascular Molecular Biology and Regulatory Peptides, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No